CLINICAL TRIAL: NCT05055544
Title: BeaRberry in the Treatment of Acute UncoMplIcated Cystitis (BRUMI)- Protocol of a Multicentre, Randomized Double-Blind Clinical Trial
Brief Title: Bearberry in the Treatment of Cystitis
Acronym: BRUMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dezső Csupor, associate professor, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IV/4225-1/2021/EKU
Record Dates: First submitted 2021-09-11; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Cystitis
Keywords: bearberry; cystitis; uncomplicated cystitis; fosfomycin
MeSH Terms: conditions — Cystitis | interventions — Fosfomycin; Emodin

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, double-blinded, two-armed multicentre trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fosfomycin (Active Comparator): a single dose of fosfomycin (3 g) powder dissolved in 75 ml water and 2 placebo tablets t.i.d. for 7 days (group A)
  Interventions: Drug: Fosfomycin
- Bearberry (Active Comparator): a single dose of placebo powder dissolved in 75 ml water and 2 bearberry tablets t.i.d. for 7 days (group B).
  Interventions: Drug: Bearberry

INTERVENTIONS:
Drug: Fosfomycin — a single dose of fosfomycin (3 g) powder dissolved in 75 ml water and 2 placebo tablets t.i.d. for 7 days (group A),
  Arms: Fosfomycin
Drug: Bearberry — a single dose of placebo powder dissolved in 75 ml water and 2 bearberry tablets t.i.d. for 7 days (group B).
  Arms: Bearberry

SUMMARY:
The goal of this study is to assess the efficacy of bearberry in uncomplicated cystitis. Uncomplicated cystitis is a disease related to the infection of the urinary bladder. Typical symptoms are dysuria, urinary urgency, and frequent voiding of small volumes. Urinary tract infections are frequent in women, usually treated with antibiotics, since the disease is usually caused by bacteria.

Fosfomycin is a frequently used antibiotic for the treatment of uncomplicated cystitis. This medicine is typically prescribed by MDs. However, since uncomplicated cystitis is quite frequent, not all patients visit the doctor when experiencing the symptoms of this disease. The use of over-the-counter products (medicines and food supplements) to alleviate the symptoms is common. One of the most frequently used medicinal plants for this purpose is bearberry. Bearberry is a medicinal plant traditionally used for the treatment of cystitis. Its use is accepted by the European Medicine Agency as traditional herbal medicinal product for relief of symptoms of mild recurrent lower urinary tract infections such as burning sensation during urination and/or frequent urination in women. Although the experience gained during the traditional use and the laboratory experiments support the supposed beneficial effect of bearberry, its clinical efficacy has not been confirmed in well-designed clinical trials in comparison with standard antibiotic therapy. In this study, the efficacy of bearberry will be assessed in comparison with fosfomycin.

Premenopausal women experiencing the symptoms of uncomplicated cystitis will be randomly divided into two groups. Since it will be a double-blind trial, neither the participants nor the experimenters will know who is receiving a particular treatment. In group A, patients will receive a single dose of fosfomycin powder dissolved in water and 2 placebo tablets three times a day for 7 days. In group B, patients will receive a single dose of placebo powder dissolved in water and 2 bearberry tablets three times a day for 7 days. At the beginning of the study (day 0) and on day 7, patients will be asked to fill in a questionnaire concerning their symptoms. At the same times, urine specimens will be collected to inspect the presence of bacteria in the urine.

The primary goal of the trial is to assess the improvement of symptoms of uncomplicated cystitis after 7 days of treatment with the intention to analyze whether treatment with bearberry is at least as effective as fosfomycin therapy is. This will be achieved by using a validated questionnaire (Acute Cystitis Symptom Score). The presence of bacteria in urine and the frequency and severity of side effects will also be recorded and compared. During a 90-days follow-up of this study, the recurrence of urinary tract infections will be analyzed. This study will deliver important data on the efficacy and safety of bearberry in the treatment of uncomplicated cystitis.

DETAILED DESCRIPTION:
This randomized, controlled double-blind multicentre trial will assess the non-inferiority of bearberry (Arctostaphylos uva-ursi) in comparison with fosfomycin in the therapy of uncomplicated cystitis.

In clinical practice, acute uncomplicated cystitis is usually treated based on the clinical signs and symptoms. According to current guidelines, first-line drugs are fosfomycin trometamol, nitrofurantoin, nitroxoline, trimethoprim-sulfamethoxazole, and pivmecillinam. The advantage of fosfomycin is that a single is considered to be sufficient for the treatment of uncomplicated cystitis, resulting in better patient compliance compared to other antibiotics.

Bacterial resistance is one of the major drawback of antibiotic use. Therefore, the assessment of other medicines than currently used antibiotics is of primary importance. One of the most widely used over-the-counter medications in the treatment of urinary tract infection-related symptoms is bearberry. Although this plant has been used in traditional medicine for the treatment of acute cystitis, and the European Medicines Agency acknowledged its use as traditional herbal medicinal product used for the treatment of symptoms of mild recurrent lower urinary tract infections such as burning sensation during urination and/or frequent urination in women, the efficacy has not been assessed in well-designed clinical trials. Since several patients are using bearberry-based medicines, it is important to obtain clinical data on the efficacy and safety of this plant. The aim of this study is to assess the non-inferiority of bearberry in comparison with a standard antibiotic (fosfomycin) used in acute uncomplicated cystitis.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal adult women
* diagnosis of acute uncomplicated cystitis (with the symptoms of dysuria, increased frequency, and urgency of urination and lower abdominal pain (suprapubic pain), that is presumed to be confined to the bladder; with no signs or symptoms that suggest an upper tract or systemic infection)
* a sum-score of of ≥6 for the typical uncomplicated urinary tract infections symptoms (frequency, urgency, painful urination, incomplete emptying, suprapubic pain, and visible hematuria) reported on the Acute Cystitis Symptom Score (ACSS) typical domain and pyuria (10 white blood cells/mm3 in a mid-stream specimen) at day 0

Exclusion Criteria:

* any renal disease
* upper urinary tract infection
* malformations of the urinary tract
* congenital disorders of the urinary tract
* catheter use
* pregnancy
* breastfeeding
* self-medication with bearberry or antibiotic use in the last 3 months
* 5 or more bearberry treatments in the previous year
* concomitant use of other antibiotics and NSAIDs
* contraindication for study drugs
* active malignancy
* immunodeficiency, including immunosuppressive treatment.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 504 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of symptom severity | The 2 time points at which the measurement is assessed is the time of enrollment, after 7 days of treatment.
  the change of symptom severity of uncomplicated cystitis after 7 days of treatment. The improvement of symptoms will be determined by using the validated Hungarian version of the Acute Cystitis Symptom Score on day 0 and day 7 according to predefined thresholds

SECONDARY OUTCOMES:
Number of patients without significant urine pathogens | The time point at which the measurement is assessed on day 7.
  number of patients with urine with <103 colony forming units (CFU)/ml on day 7
Number of urine pathogens | The time point at which the measurement is assessed on day 7.
  average number of CFU of pathogens (7 days after the start of the therapy) in urine
Frequency and severity of side effects | The time point at which the measurement is assessed on day 7.
  frequency and severity of side effects used a questionnaire
Recurrence of urinary tract infection (UTI) | The time point at which the measurement is assessed on day 90.
  follow-up after 90 days; severity and diagnostics of recurrences to be assessed by using the ACSS
Concurrent use of other medications | The time point at which the measurement is assessed on day 7.
  concurrent use of other over-the-counter (OTC) medications and food supplements that are started taking during the 7 day treatment trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
URL: http://tm-centre.org/

REFERENCES:
- [Background] Naber KG, Schito G, Botto H, Palou J, Mazzei T. Surveillance study in Europe and Brazil on clinical aspects and Antimicrobial Resistance Epidemiology in Females with Cystitis (ARESC): implications for empiric therapy. Eur Urol. 2008 Nov;54(5):1164-75. doi: 10.1016/j.eururo.2008.05.010. Epub 2008 May 21. PMID 18511178
- [Background] Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, Moran GJ, Nicolle LE, Raz R, Schaeffer AJ, Soper DE; Infectious Diseases Society of America; European Society for Microbiology and Infectious Diseases. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: A 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011 Mar 1;52(5):e103-20. doi: 10.1093/cid/ciq257. PMID 21292654
- [Background] Keating GM. Fosfomycin trometamol: a review of its use as a single-dose oral treatment for patients with acute lower urinary tract infections and pregnant women with asymptomatic bacteriuria. Drugs. 2013 Nov;73(17):1951-66. doi: 10.1007/s40265-013-0143-y. PMID 24202878
- [Background] Schmiemann G, Kniehl E, Gebhardt K, Matejczyk MM, Hummers-Pradier E. The diagnosis of urinary tract infection: a systematic review. Dtsch Arztebl Int. 2010 May;107(21):361-7. doi: 10.3238/arztebl.2010.0361. Epub 2010 May 28. PMID 20539810
- [Background] Kranz J, Schmidt S, Lebert C, Schneidewind L, Mandraka F, Kunze M, Helbig S, Vahlensieck W, Naber K, Schmiemann G, Wagenlehner FM. The 2017 Update of the German Clinical Guideline on Epidemiology, Diagnostics, Therapy, Prevention, and Management of Uncomplicated Urinary Tract Infections in Adult Patients. Part II: Therapy and Prevention. Urol Int. 2018;100(3):271-278. doi: 10.1159/000487645. Epub 2018 Mar 14. PMID 29539622
- [Background] Gardiner BJ, Stewardson AJ, Abbott IJ, Peleg AY. Nitrofurantoin and fosfomycin for resistant urinary tract infections: old drugs for emerging problems. Aust Prescr. 2019 Feb;42(1):14-19. doi: 10.18773/austprescr.2019.002. Epub 2019 Feb 1. PMID 30765904
- [Background] Falagas ME, Vouloumanou EK, Samonis G, Vardakas KZ. Fosfomycin. Clin Microbiol Rev. 2016 Apr;29(2):321-47. doi: 10.1128/CMR.00068-15. PMID 26960938
- [Background] Van Pienbroek E, Hermans J, Kaptein AA, Mulder JD. Fosfomycin trometamol in a single dose versus seven days nitrofurantoin in the treatment of acute uncomplicated urinary tract infections in women. Pharm World Sci. 1993 Dec 17;15(6):257-62. doi: 10.1007/BF01871127. PMID 8298585
- [Background] Stein GE. Comparison of single-dose fosfomycin and a 7-day course of nitrofurantoin in female patients with uncomplicated urinary tract infection. Clin Ther. 1999 Nov;21(11):1864-72. doi: 10.1016/S0149-2918(00)86734-X. PMID 10890258
- [Background] Minassian MA, Lewis DA, Chattopadhyay D, Bovill B, Duckworth GJ, Williams JD. A comparison between single-dose fosfomycin trometamol (Monuril) and a 5-day course of trimethoprim in the treatment of uncomplicated lower urinary tract infection in women. Int J Antimicrob Agents. 1998 Apr;10(1):39-47. doi: 10.1016/s0924-8579(98)00021-1. PMID 9624542
- [Background] Huttner A, Kowalczyk A, Turjeman A, Babich T, Brossier C, Eliakim-Raz N, Kosiek K, Martinez de Tejada B, Roux X, Shiber S, Theuretzbacher U, von Dach E, Yahav D, Leibovici L, Godycki-Cwirko M, Mouton JW, Harbarth S. Effect of 5-Day Nitrofurantoin vs Single-Dose Fosfomycin on Clinical Resolution of Uncomplicated Lower Urinary Tract Infection in Women: A Randomized Clinical Trial. JAMA. 2018 May 1;319(17):1781-1789. doi: 10.1001/jama.2018.3627. PMID 29710295
- [Background] Loras C, Mendes AC, Peixe L, Novais A, Alos JI. Escherichia coli resistant to fosfomycin from urinary tract infections: Detection of the fosA3 gene in Spain. J Glob Antimicrob Resist. 2020 Jun;21:414-416. doi: 10.1016/j.jgar.2020.01.023. Epub 2020 Feb 12. PMID 32061811
- [Background] Oteo J, Bautista V, Lara N, Cuevas O, Arroyo M, Fernandez S, Lazaro E, de Abajo FJ, Campos J; Spanish ESBL-EARS-Net Study Group. Parallel increase in community use of fosfomycin and resistance to fosfomycin in extended-spectrum beta-lactamase (ESBL)-producing Escherichia coli. J Antimicrob Chemother. 2010 Nov;65(11):2459-63. doi: 10.1093/jac/dkq346. Epub 2010 Sep 16. PMID 20851815
- [Background] Moskalenko SA. Preliminary screening of far-eastern ethnomedicinal plants for antibacterial activity. J Ethnopharmacol. 1986 Mar;15(3):231-59. doi: 10.1016/0378-8741(86)90163-7. PMID 3724205
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Jahodar L, Leifertova I, Lisa M. Elimination of arbutin from the organism. Pharmazie. 1983 Nov;38(11):780-1. No abstract available. PMID 6669604
- [Background] Divincenzo GD, Hamilton ML, Reynolds RC, Ziegler DA. Metabolic fate and disposition of [14C]hydroquinone given orally to Sprague-Dawley rats. Toxicology. 1984 Oct;33(1):9-18. doi: 10.1016/0300-483x(84)90012-x. PMID 6495348
- [Background] Glockl I, Blaschke G, Vei M. Validated methods for direct determination of hydroquinone glucuronide and sulfate in human urine after oral intake of bearberry leaf extract by capillary zone electrophoresis. J Chromatogr B Biomed Sci Appl. 2001 Sep 25;761(2):261-6. doi: 10.1016/s0378-4347(01)00322-x. PMID 11587357
- [Background] Alidjanov JF, Abdufattaev UA, Makhsudov SA, Pilatz A, Akilov FA, Naber KG, Wagenlehner FM. New self-reporting questionnaire to assess urinary tract infections and differential diagnosis: acute cystitis symptom score. Urol Int. 2014;92(2):230-6. doi: 10.1159/000356177. Epub 2014 Jan 23. PMID 24457349
- [Background] Magyar A, Alidjanov J, Pilatz A, Nagy K, Arthanareeswaran VKA, Poth S, Becsi A, Wagenlehner FME, Naber KG, Tenke P, Koves B. The role of the Acute Cystitis Symptom Score questionnaire for research and antimicrobial stewardship. Validation of the Hungarian version. Cent European J Urol. 2018;71(1):134-141. doi: 10.5173/ceju.2018.1530. Epub 2017 Jan 22. PMID 29732220
- [Derived] Toth B, Javorhazy A, Nyirady P, Csupor-Loffler B, Birinyi P, Zhanel G, Naber K, Langer R, Vorhendi N, Gede N, Vancsa S, Hegyi P, Csupor D. Bearberry in the treatment of acute uncomplicated cystitis (BRUMI): protocol of a multicentre, randomised double-blind clinical trial. BMJ Open. 2022 Jun 24;12(6):e057982. doi: 10.1136/bmjopen-2021-057982. PMID 35750460
- See also: Related Info — http://tm-centre.org/